CLINICAL TRIAL: NCT02790567
Title: Evaluation of Automated Immunoassay, Particle Gel Immunoassay and Pretest Scoring Systems (4Ts and HEP Scores) in the Diagnosis of Heparin-induced Thrombocytopenia in Surgical Critically Ill Patients
Brief Title: Rapid Diagnosis of Heparin-Induced Thrombocytopenia in Surgical Critically Ill Patients
Acronym: TIH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: TIH-2012
Record Dates: First submitted 2013-08-01; First posted 2016-06-06 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2013-05

CONDITIONS: Heparin-induced Thrombocytopenia (HIT)
Keywords: diagnostic performance; heparin-induced thrombocytopenia; rapid immunological diagnostic method; immunoassay; pretest scoring systems; 4Ts score; HEP score
MeSH Terms: interventions — Latex Fixation Tests

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIT study group: The HIT study group will include all patients admitted in our surgical intensive care unit (ICU) during the study period if the clinician in charge of the patient suspects the diagnosis of HIT. The HEP score, the 4Ts score, the immuno-diffusion particle gel immunoassay (ID-PaGIA) and the HIT-Ab(PF4-H) test will be done for each patient the day the diagnosis of HIT will be suspected.
  Interventions: Other: HEP score; Other: 4Ts score; Other: ID-PaGIA test; Other: HIT-Ab(PF4-H) test

INTERVENTIONS:
Other: HEP score — The HEP score is a clinicobiological score evaluating the probability of the HIT diagnosis.
  The HEP score is based on the blood platelet count, the timing of the platelet decrease, the existence of clinical manifestations of HIT (thrombosis, haemorrhage, skin necrosis) and the existence of an other cause of thrombocytopenia.
  Other Names: The HEP score is the HIT Expert Probability score.
Other: 4Ts score — The 4Ts score is a clinicobiological score evaluating the probability of the HIT diagnosis. The 4Ts score is based on the change in blood platelet count during heparin therapy, the timing of platelet decrease, the existence of a thrombosis, and the existence of an other cause of thrombocytopenia.
Other: ID-PaGIA test — The ID-PaGIA test is a particle gel immunoassay that detects immunoglobulins (Ig) G, A and M specific to the heparin/PF4 complexes.
Other: HIT-Ab(PF4-H) test — The HIT-Ab(PF4-H) test consist in the incubation of plasma samples with latex beads coated PF4/polyvinylsulfate complexes. After binding of the plasma antibodies a monoclonal antibody recognizing PF4/heparin complexes is added. In the presence of human anti-PF4/heparin antibodies, binding of the monoclonal antibody and subsequent agglutination of latex beads is inhibited. Inhibition of agglutination is quantified and reported in arbitrary units (U/ml). A value equal or higher than 1.0 u/ml may indicate the presence of HIT antibodies.
  Other Names: HIT-Ab(PF4-H) latex agglutination test

SUMMARY:
The early diagnosis of heparin-induced thrombocytopenia is particularly difficult in surgical critically ill patients. If the use of rapid immunological diagnostic methods and pretest scoring systems has been proposed in the medical intensive care unit (ICU), none of these methods have been specifically evaluated in the diagnosis of HIT in surgical patients.

DETAILED DESCRIPTION:
Heparin-induced thrombocytopenia (HIT) is of concern in critically ill patients, given the high prevalence of heparin use. The diagnosis of HIT in surgical intensive care unit (ICU) is problematic due to the lack of reliable diagnostic method. No gold standard currently exists and the definitive diagnosis is mainly based on the detection of heparin-dependent platelet-activating antibodies by ELISA method, on the platelet serotonin release assay (SRA) and on the changes of the blood platelet count after the discontinuation of heparin therapy. As a result, no early definitive diagnosis could be done. This could expose patients to thrombotic complications related to the HIT or hemorrhagic complications related to the alternative anticoagulant prescribed. This complications can threaten the prognosis of these patients. Particle gel immunoassay and automated immunoassay has been proposed for the early diagnosis of HIT in medical critically ill and non-critically ill patients. Many authors suggest that the accuracy of these immunological methods for the diagnosis of HIT could be altered in surgical patients, but these tests has never been specifically evaluated in this population. The 4Ts and the HIT Expert Probability (HEP) score systems sound interesting for the diagnosis of HIT. These clinicobiological scores can be easily used by non-expert clinicians, but have also never been evaluated in the surgical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosis of HIT suspected
* Admitted in our surgical intensive care unit during the study period

Exclusion Criteria:

* Age < 18 years old
* Pregnancy and/or breast feeding
* Fondaparinux anticoagulation
* Withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in our surgical intensive care unit (ICU) during the study period will be elligible if the diagnosis of HIT is supected by the attending physician. The diagnosis of the HIT will be suspected in the presence of at least one of the following criteria in a patient receiving an heparin therapy: (1) a thrombocytopenia < 100 G/l or a decrease of the blood platelet count > 40%, (2) a thrombocytopenia between the 5th and the 8th of the heparin therapy, (3)an arterial or a venous thrombosis in a patient receiving heparin, (4)the failure of a treatment of a thrombosis with heparin. These criteria are described in the French guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sensibility, specificity, positive and negative predictive values of HEP score for the diagnosis of heparin-induced thrombocytopenia (HIT) | during the ICU stay, i.e an average time of 10 days

SECONDARY OUTCOMES:
Sensibility, specificity, positive and negative predictive values of the 4Ts score for the diagnosis of heparin-induced thrombocytopenia (HIT) | during the ICU stay, i.e an average time of 10 days
  Sensibility, specificity, positive and negative predictive values of the 4Ts score for the diagnosis of heparin-induced thrombocytopenia (HIT)
Sensibility, specificity, positive and negative predictive value of the particul gel immunoassay ID-PaGia test for the diagnosis of heparin-induced thrombocytopenia (HIT) | during the ICU stay, i.e an average time of 10 days
  Sensibility, specificity, positive and negative predictive value of the particul gel immunoassay ID-PaGia test for the diagnosis of heparin-induced thrombocytopenia (HIT)
Sensibility, specificity, positive and negative predictive values of the automated immunoassay HemosIL-Ab latex agglutination test for the diagnosis of heparin-induced thrombocytopenia (HIT) | during the ICU stay, i.e an average time of 10 days
  Sensibility, specificity, positive and negative predictive values of the automated immunoassay HemosIL-Ab latex agglutination test for the diagnosis of heparin-induced thrombocytopenia (HIT)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ginet, MD, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France